CLINICAL TRIAL: NCT03982680
Title: Clinical Study of Toripalimab Monoclonal Antibody Combined With Gemcitabine/5--fluoropyrimidine in the Treatment of Advanced Cholangiocarcinoma
Brief Title: Toripalimab Combined With Gemcitabine/5--fluoropyrimidine for Advanced Cholangiocarcinoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Jiangmen Central Hospital (Other)
Responsible Party: Principal Investigator, yu gengsheng, Vice director of Oncology department, Jiangmen Central Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: cholangiocarcinoma
Record Dates: First submitted 2019-06-07; First posted 2019-06-11 (Actual); Last update posted 2019-07-16 (Actual); Status verified 2019-07

CONDITIONS: Advanced Cholangiocarcinoma
MeSH Terms: interventions — toripalimab; Gemcitabine; Fluorouracil

STUDY DESIGN:
Intervention Model Description: All patients were given Toripalimab 3 mg/kg (day 1 and 15); Gem+5-FU (Gem 1250mg/m2+CF 200 mg/m2+5-FU400 mg/m2 intravenous drip+5-FU 2.4-3.6 g/m2 continuous intravenous drip for 48 hours), the first and fifteenth days, four weeks for a cycle, a total of four cycles. After 4 cycles, Toripalimab was maintained at 3 mg/kg Q3 w for a total of 1 year if the disease was not progressing or toxic side effects were tolerated.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Toripalimab combined with Gem/5-FU (Experimental): All patients were given Toripalimab 3 mg/kg (day 1 and 15); Gem+5-FU (Gem 1250mg/m2+CF 200 mg/m2+5-FU400 mg/m2 intravenous drip+5-FU 2.4-3.6 g/m2 continuous intravenous drip for 48 hours), the first and fifteenth days, four weeks for a cycle, a total of four cycles.After 4 cycles, Toripalimab was maintained at 3 mg/kg Q3 w for a total of 1 year if the disease was not progressing or toxic side effects were tolerated.
  Interventions: Drug: Toripalimab; Drug: Gemcitabine; Drug: 5- fluorine pyrimidine

INTERVENTIONS:
Drug: Toripalimab — 3mg/kg on d1 and d15 q4W*4cycles，then 3mg/kg q3w for 1 year in total
Drug: Gemcitabine — 1250mg/m2 on d1 and d15 q4W*4cycles
  Other Names: Gem
Drug: 5- fluorine pyrimidine — 400mg/m2 intravenous injection plus 5-FU 2.4g-3.6g/m2 continuous intravenous drip for 48h on d1 and d15 q4W*4cycles
  Other Names: 5-FU

SUMMARY:
The study is a phase II clinical trial of single arm. The purpose is to evaluate the safety and efficacy of anti-PD-1 antibody Toripalimab combined with chemotherapy(gemcitabine+5-fluorine pyrimidine) in unresectable advanced cholangiocarcinoma patients.

ELIGIBILITY:
Inclusion Criteria:

* histologically or cytologically confirmed cholangiocarcinoma
* stage IV disease,no system therapy for advanced disease
* one or more lesions that can be measured by imaging assessment
* 18 to 70 years of age and life expectancy exceeds 3 months
* adequate specimens for detection of PD-1/PD-L1 and MMR
* karnofsky performance status(KPS) score ≥70%
* routine blood routine, liver and kidney function and electrocardiogram were basically normal without contraindication of chemotherapy.

Exclusion Criteria:

* dual cancers other than cholangiocarcinoma
* metastasis of central nervous system
* unreleased biliary obstruction
* acute infections requiring treatment
* non-infectious pneumonia requires glucocorticoid therapy, active autoimmune diseases, or systemic immunosuppressive therapy.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2019-07-13 (Actual); Primary Completion 2021-05-30 (Estimated); Study Completion 2021-12-30 (Estimated)

PRIMARY OUTCOMES:
6-month PFS rate | 6-month after the beginning of first line systemic therapy
  the rate of 6-month progression free survival
mPFS | from the beginning of the first line systemic therapy until the date of first documented progression or date of death from any cause,whichever came first,assessed up to 24 months
  the median of progression free survival
Toxic side effects | from the beginning of the first line systemic therapy until the end of follow-up,assessed up to 24 months
  assess according to the National Cancer Institute-Common Terminology Criteria for Adverse Events 3.0

SECONDARY OUTCOMES:
ORR | from the beginning of the first line systemic therapy until the date of completion of therapy,assessed up to 13 months
  the objective response rate
DCR | from the beginning of the first line systemic therapy until the date of completion of therapy,assessed up to 13 months
  the disease control rate
1-year OS rate | 1 year after the beginning of the first line systemic therapy
  the rate of 1-year overall survival
mOS | from the beginning of the first line systemic therapy until the date of death from any cause,assessed up to 24 months
  the median of overall survival

OTHER OUTCOMES:
the value of PD-1/PD-L1 | from the beginning of the first line systemic therapy until the end of follow-up,assessed up to 24 months
  to analyze the predictive value of PD-1/PD-L1 for efficacy and toxicity
the value of MMR | from the beginning of the first line systemic therapy until the end of follow-up,assessed up to 24 months
  to analyze the predictive value of MMR for efficacy and toxicity

CONTACTS AND LOCATIONS:
Overall Officials: Yu gengsheng, master, Study Director — jiangmen cenctral hospital
Locations (1):
- Jiangmen central hospital, Jiangmen, Guangdong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] GBD 2013 Mortality and Causes of Death Collaborators. Global, regional, and national age-sex specific all-cause and cause-specific mortality for 240 causes of death, 1990-2013: a systematic analysis for the Global Burden of Disease Study 2013. Lancet. 2015 Jan 10;385(9963):117-71. doi: 10.1016/S0140-6736(14)61682-2. Epub 2014 Dec 18. PMID 25530442
- [Background] Jain A, Javle M. Molecular profiling of biliary tract cancer: a target rich disease. J Gastrointest Oncol. 2016 Oct;7(5):797-803. doi: 10.21037/jgo.2016.09.01. PMID 27747093
- [Background] Takakura H, Domae S, Ono T, Sasaki A. The Immunological Impact of Chemotherapy on the Tumor Microenvironment of Oral Squamous Cell Carcinoma. Acta Med Okayama. 2017 Jun;71(3):219-226. doi: 10.18926/AMO/55204. PMID 28655941
- [Background] Gotwals P, Cameron S, Cipolletta D, Cremasco V, Crystal A, Hewes B, Mueller B, Quaratino S, Sabatos-Peyton C, Petruzzelli L, Engelman JA, Dranoff G. Prospects for combining targeted and conventional cancer therapy with immunotherapy. Nat Rev Cancer. 2017 May;17(5):286-301. doi: 10.1038/nrc.2017.17. Epub 2017 Mar 24. PMID 28338065
- [Background] Okusaka T, Nakachi K, Fukutomi A, Mizuno N, Ohkawa S, Funakoshi A, Nagino M, Kondo S, Nagaoka S, Funai J, Koshiji M, Nambu Y, Furuse J, Miyazaki M, Nimura Y. Gemcitabine alone or in combination with cisplatin in patients with biliary tract cancer: a comparative multicentre study in Japan. Br J Cancer. 2010 Aug 10;103(4):469-74. doi: 10.1038/sj.bjc.6605779. Epub 2010 Jul 13. PMID 20628385
- [Background] Morizane C, Ueno M, Ikeda M, Okusaka T, Ishii H, Furuse J. New developments in systemic therapy for advanced biliary tract cancer. Jpn J Clin Oncol. 2018 Aug 1;48(8):703-711. doi: 10.1093/jjco/hyy082. PMID 29893894
- [Background] Sabbatino F, Villani V, Yearley JH, Deshpande V, Cai L, Konstantinidis IT, Moon C, Nota S, Wang Y, Al-Sukaini A, Zhu AX, Goyal L, Ting DT, Bardeesy N, Hong TS, Fernandez-del Castillo C, Tanabe KK, Lillemoe KD, Ferrone S, Ferrone CR. PD-L1 and HLA Class I Antigen Expression and Clinical Course of the Disease in Intrahepatic Cholangiocarcinoma. Clin Cancer Res. 2016 Jan 15;22(2):470-8. doi: 10.1158/1078-0432.CCR-15-0715. Epub 2015 Sep 15. PMID 26373575
- [Background] Taube JM, Klein A, Brahmer JR, Xu H, Pan X, Kim JH, Chen L, Pardoll DM, Topalian SL, Anders RA. Association of PD-1, PD-1 ligands, and other features of the tumor immune microenvironment with response to anti-PD-1 therapy. Clin Cancer Res. 2014 Oct 1;20(19):5064-74. doi: 10.1158/1078-0432.CCR-13-3271. Epub 2014 Apr 8. PMID 24714771
- [Background] Herbst RS, Soria JC, Kowanetz M, Fine GD, Hamid O, Gordon MS, Sosman JA, McDermott DF, Powderly JD, Gettinger SN, Kohrt HE, Horn L, Lawrence DP, Rost S, Leabman M, Xiao Y, Mokatrin A, Koeppen H, Hegde PS, Mellman I, Chen DS, Hodi FS. Predictive correlates of response to the anti-PD-L1 antibody MPDL3280A in cancer patients. Nature. 2014 Nov 27;515(7528):563-7. doi: 10.1038/nature14011. PMID 25428504
- [Background] Topalian SL, Hodi FS, Brahmer JR, Gettinger SN, Smith DC, McDermott DF, Powderly JD, Carvajal RD, Sosman JA, Atkins MB, Leming PD, Spigel DR, Antonia SJ, Horn L, Drake CG, Pardoll DM, Chen L, Sharfman WH, Anders RA, Taube JM, McMiller TL, Xu H, Korman AJ, Jure-Kunkel M, Agrawal S, McDonald D, Kollia GD, Gupta A, Wigginton JM, Sznol M. Safety, activity, and immune correlates of anti-PD-1 antibody in cancer. N Engl J Med. 2012 Jun 28;366(26):2443-54. doi: 10.1056/NEJMoa1200690. Epub 2012 Jun 2. PMID 22658127
- [Background] Gou M, Zhang Y, Si H, Dai G. Efficacy and safety of nivolumab for metastatic biliary tract cancer. Onco Targets Ther. 2019 Jan 25;12:861-867. doi: 10.2147/OTT.S195537. eCollection 2019. PMID 30774373
- [Background] Asaoka Y, Ijichi H, Koike K. PD-1 Blockade in Tumors with Mismatch-Repair Deficiency. N Engl J Med. 2015 Nov 12;373(20):1979. doi: 10.1056/NEJMc1510353. No abstract available. PMID 26559583